CLINICAL TRIAL: NCT06924229
Title: Corneal Changes in Estrogen-Dependent Breast Cancer After Hormonal Treatment
Acronym: breast cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Haitham Thabit, Dr., Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-24-03-14PD
Record Dates: First submitted 2025-03-17; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-06

CONDITIONS: Braest Cancer; Dry Eye
Keywords: corneal changes; breast cancer; hormonal treatment
MeSH Terms: conditions — Dry Eye Syndromes; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patients with breast cancer recieving hormonal treatment (Active Comparator): evaluation of the effect of hormonal treatment on the cornea
  Interventions: Drug: Hormonal treatment

INTERVENTIONS:
Drug: Hormonal treatment — hormonal treatment for breast cancer

SUMMARY:
Aromatase inhibitors (AI) therapy is the treatment of choice for estrogen receptor-positive breast cancer (BC). While AIs effectively suppress tumor growth, estrogen deprivation may have negative impacts on the eyes. This work evaluated the anterior segment changes in estrogen-dependent BC after hormonal treatment.

DETAILED DESCRIPTION:
Aromatase inhibitors (AI) therapy is an important treatment for estrogen receptor-positive breast cancer (BC). This work evaluated the eye anterior segment changes in estrogen-dependent BC after hormonal treatment.

This cross-sectional study was conducted on female patients aged ≥18 who received treatment for BC. Patients were evaluated by a number of tests to determine the effects on the cornea and the lacrimal system

ELIGIBILITY:
Inclusion Criteria:

* Females diagnosed with breast cancer

Exclusion Criteria:

* uncontrolled diabetes , auto immune diseases

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
tear break up time test and shirmer test | 6 months
  these tests done before starting treatment and in follow up after recieving treatment to evaluate the lacrimal function and dry eye

SECONDARY OUTCOMES:
Corneal thickness and endothelium hexagonality | 6 months
  Corneal thickness and hesagonality were evaluated before and after treatment with aromatase inhibitors

CONTACTS AND LOCATIONS:
Overall Officials: Elshimaa abd almateen A mateen, Doctorate, Study Chair — Sohag University; alaa mahmoud m mahmoud, Study Chair — mahmoud; mohamed salah hamed s hamed, Doctorate, Study Director — Sohag University
Locations (1):
- Sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: breast cancer therapy — https://link.springer.com/chapter/10.1007/978-3-031-70875-6_22